CLINICAL TRIAL: NCT01910350
Title: Kin KeeperSM: Reducing Disparities Through Cancer Literacy and Screening
Acronym: KinKeeper
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Michigan State University (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Principal Investigator, Karen Williams, Professor, Michigan State University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 10-256; 1R01NR011323 (NIH)
Record Dates: First submitted 2013-07-25; First posted 2013-07-29 (Estimated); Last update posted 2015-09-25 (Estimated); Status verified 2015-09

CONDITIONS: Breast Cancer; Cervical Cancer
Keywords: Breast & cervical cancer prevention & screening
MeSH Terms: conditions — Breast Neoplasms; Uterine Cervical Neoplasms | interventions — Standard of Care

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cancer prevention intervention (Experimental): Cancer prevention intervention: Experimental group receives intensive 2 hour education in each breast and cervical cancer risks and prevention intervention, and face to face reading of post intervention surveys by an community health worker.
  Interventions: Behavioral: Kin KeeperSM Cancer Prevention Intervention
- Control group receives standard care (Active Comparator): The control group receives reading materials and brochures on breast and cervical cancer such as one would receive in a doctors office and post condition surveys. All materials are read by the participant without the interaction or assistance of the community health worker.
  Interventions: Other: Standard of care

INTERVENTIONS:
Behavioral: Kin KeeperSM Cancer Prevention Intervention
  Arms: Cancer prevention intervention
Other: Standard of care
  Arms: Control group receives standard care

SUMMARY:
1) To determine if the Kin KeeperSM Cancer Prevention Intervention increases first time and appropriately timed breast cancer screening rates among Black, Latina and Arab women; 2) To determine if the Kin KeeperSM Cancer Prevention Intervention increase first time and appropriately time cervical cancer screening rates among Black, Latina and Arab women; 3) To measure functional cancer literacy over time at the individual and familial level and 4) Assess rates of healthcare utilization cost among women in the Kin KeeperSM intervention and control-comparison groups.

ELIGIBILITY:
Inclusion Criteria:

* Participants:self-identified as Black Latina and Arab women ho can recruit at least two bloodline female family members (mother daughter sister, etc.; can accommodate two in-home visits by a community health worker; and 21-70 years of age.

Exclusion Criteria:

* are not self-identified as Black, Latina, or Arab; do not have direct bloodline relatives; and are younger than 21 or older than 70 years of age.

Ages: 21 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 516 (Actual)
Dates: Start 2010-07; Primary Completion 2015-02 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
First time AND appropriately timed, clinical breast exam, mammogram, pap test | Baseline through 36 months.
  Participants will complete measures every 6 months (baseline, 12 mo., 18 mo., 24 mo., 30 mo. & 36 mo.)to measure increases in screening rates for experimental vs. control group.

SECONDARY OUTCOMES:
Increased Breast and Cervical Cancer Literacy rates. | Baseline-36 months.
  Do participants have a higher breast and cervical cancer literacy rates post intervention and over 36 months than control group as well as better retention?

CONTACTS AND LOCATIONS:
Locations (1):
- Michigan State University, East Lansing, Michigan, United States

REFERENCES:
- [Background] Williams KP, Roman L, Meghea CI, Penner L, Hammad A, Gardiner J. Kin KeeperSM: design and baseline characteristics of a community-based randomized controlled trial promoting cancer screening in Black, Latina, and Arab women. Contemp Clin Trials. 2013 Mar;34(2):312-9. doi: 10.1016/j.cct.2012.12.005. Epub 2012 Dec 28. PMID 23274402